CLINICAL TRIAL: NCT01496690
Title: Pregablin for Anxiety-comorbidity in Patients With Schizophrenia - a Double-blinded Randomized Placebo Controlled Study
Brief Title: Pregablin for Anxiety-comorbidity in Patients With Schizophrenia
Acronym: PACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Albert Einstein College of Medicine (Other); GCP-unit at Aarhus University Hospital, Aarhus, Denmark (Other); The Hospital Pharmcacy North Denmark Region, Denmark (Unknown); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Eudra CT nr 2010-024488-42; N-20100097 (Other: The North Denmark Region Committee on Health Research Ethics)
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Schizophrenia; Anxiety-comorbidity to Schizophrenia
Keywords: Anxiety-comorbidity to schizophrenia; Double-blinded randomized placebo controlled trial; Pregabalin
MeSH Terms: conditions — Schizophrenia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pregabalin (Active Comparator): The pregabalin dose is 75 mg daily the first week followed by 7 weeks of flexible daily dosing (150, 300, 450 or 600 mg.) depending on tolerability and response.
  Interventions: Drug: Pregabalin
- Pregabalin Placebo Capsules (Placebo Comparator)
  Interventions: Drug: Pregabalin Placebo Capsules

INTERVENTIONS:
Drug: Pregabalin — Subjects are randomized 1:1 to either pregabalin treatment or placebo. The intervention period is 8 weeks. The daily pregabalin dose is 75 mg. during the first week followed by 7 weeks of flexible daily dosing (150, 300, 450 or 600 mg.) depending on tolerability and response. Doses above 150 mg. should be divided in two daily dosages.
  Other Names: Brand name: Lyrica(R)
  Arms: pregabalin
Drug: Pregabalin Placebo Capsules — Parallel to Active Comparator
  Arms: Pregabalin Placebo Capsules

SUMMARY:
The PACS study aims to investigate the efficacy and tolerability of pregabalin for schizophrenic patients that suffer from comorbid anxiety.

The study design is an 8 week flexible dosage, randomized placebo controlled.

The study population is patients diagnosed with ICD-10 schizophrenia and age 18-65. Patients are recruited from outpatient clinics from entire Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years
* An ICD-10 schizophrenia diagnosis F20.0-20.3 or F20.9
* Stable dosage of psychotropic 4 weeks before inclusion
* Hamilton Anxiety Scale total score > 15
* Positive and Negative Syndrome Scale for Schizophrenia total score < 70
* The Calgary Depression Scale for Schizophrenia total score < 10
* Fertile women: Contraception during the trial
* S-creatinin within normal reference range
* Signed informed consent and power of attorney

Exclusion Criteria:

* Significant substance abuse
* QTc > 480 milliseconds
* Severe dysregulated diabetes
* For women: Pregnancy or breast-feeding
* Confinement in accordance with the Danish Law of Psychiatry
* Concrete suicidally
* Known hypersensitivity or allergic reaction to the active ingredient of the drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale | Baseline - 4 weeks treatment - 8 weeks treatment

SECONDARY OUTCOMES:
UKU-Overall adverse effect scale | Baseline - 4 weeks treatment - 8 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ole Schjerning, M.D., Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Psychiatry, Aalborg, Denmark